CLINICAL TRIAL: NCT05983159
Title: A Modular Open Label, Signal Seeking, Phase II Trial of Targeted Therapies for Patients With Slow-Flow or Fast-Flow Vascular Malformations (TARGET-VM)
Brief Title: A Trial of Targeted Therapies for Patients With Slow-Flow or Fast-Flow Vascular Malformations
Acronym: TARGET-VM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other); Royal Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 85218
Record Dates: First submitted 2023-07-27; First posted 2023-08-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Slow-Flow Vascular Malformation; Fast-Flow Vascular Malformation; Vascular Malformations; Venous Malformation; Lymphatic Malformation, Low Flow; Lymphatic Malformation; Lymphangioma; Arteriovenous Malformations; Venous Malformation, Low Flow; Cystic Hygroma; Vascular Anomaly; Vascular Anomalies; PI3K Gene Mutation; MAP2K1 Gene Mutation; PIK3CA-related Overgrowth Spectrum; Arteriovenous Malformation (AVM); KRAS G12C; KRAS G12D
Keywords: Targeted therapy; vascular malformations; skin diseases, vascular; Phosphatidylinositol 3-Kinases; MEK inhibitor 1
MeSH Terms: conditions — Vascular Malformations; Lymphatic Abnormalities; Lymphangioma; Arteriovenous Malformations; Lymphangioma, Cystic; Skin Diseases, Vascular | interventions — Alpelisib; mirdametinib

STUDY DESIGN:
Intervention Model Description: i) Participants with slow-flow vascular malformations with an eligible gene mutation will receive 48 weeks of treatment with open-label alpelisib.
  ii) Participants with fast-flow vascular malformations with an eligible gene mutation will receive 48 weeks of treatment with open-label mirdametinib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Module 1: Slow-flow vascular malformations (Experimental): Slow-flow vascular malformations with identified causative variants in the phosphoinositide 3-kinase (PI3K) signalling pathway will receive alpelisib (provided by Novartis Pharmaceuticals), an oral alpha-specific PI3-kinase inhibitor for a total duration of 48 weeks as monotherapy, followed by 24 weeks of follow-up.
  Interventions: Drug: Alpelisib
- Module 2: Fast-flow vascular malformations (Experimental): Fast-flow vascular malformations with identified causative variants in the RAS-MEK-ERK signalling pathway will receive mirdametinib (provided by SpringWorks Therapeutics, Inc.), an investigational oral MEK inhibitor for a total duration of 48 weeks as monotherapy, followed by 24 weeks of follow-up.
  Interventions: Drug: Mirdametinib

INTERVENTIONS:
Drug: Alpelisib — Oral alpha-specific PI3-kinase inhibitor
  Other Names: BYL719
  Arms: Module 1: Slow-flow vascular malformations
Drug: Mirdametinib — An investigational oral MEK inhibitor
  Arms: Module 2: Fast-flow vascular malformations

SUMMARY:
Recent studies have demonstrated that growth of vascular malformations can be driven by genetic variants in one of 2 signalling pathways. Targeted drugs specific to these pathways have been developed and shown to be effective in treating cancer. This study will describe the effectiveness of (i) 48 weeks of alpelisib therapy for participants with slow-flow vascular malformations and a gene mutation in one of these signalling pathways (module 1) and (ii) 48 weeks of mirdametinib therapy for participants with fast-flow vascular malformations and a gene mutations in the other signalling pathway (module 2).

DETAILED DESCRIPTION:
TARGET-VM is a modular open-label, signal seeking, phase II trial of targeted therapies for patients with vascular malformations. Patients with vascular malformations which are refractory to standard therapies, or in whom standard therapy is not appropriate, are potentially eligible for the clinical trial. Vascular malformations will be classified as slow-flow or fast-flow lesions using established clinical criteria. Genetic testing to identify causative variants in genes affecting the phosphoinositide 3-kinase (PI3K) signalling pathway for slow-flow vascular malformations or the Mitogen-Activated Protein Kinase (MAPK) signalling pathway for fast-flow vascular malformations must be performed using research protocols or commercial testing assays that are external to this clinical trial.

The study consists of individual modules, each evaluating the clinical efficacy of 48 weeks of targeted therapy. The treatment modules are:

1. Module 1 - Treatment for slow-flow vascular malformations Eligible patients with slow-flow vascular malformations with an identified causative variant in the PI3K signalling pathway will receive alpelisib, an oral alpha-specific PI3-kinase inhibitor for a total duration of 48 weeks as monotherapy (treatment period), followed by 24 weeks of follow-up (follow-up period).
2. Module 2 - Treatment for fast-flow vascular malformations Eligible patients with fast-flow vascular malformations with an identified causative variant in the MAPK signalling pathway will receive mirdametinib, an investigational oral MEK inhibitor for a total duration of 48 weeks as monotherapy (treatment period), followed by 24 weeks of follow-up (follow-up period).

TARGET-VM will be conducted only in Victoria, Australia.

ELIGIBILITY:
MODULE 1

Inclusion Criteria:

1. Adult or paediatric patient, 2 years of age or over
2. Patient has a clinical diagnosis of a slow-flow vascular malformation
3. Patient has received standard therapy for the vascular malformation or in which, in the opinion of the investigator, standard therapy is not appropriate

   - Note: standard therapy may include treatment with sirolimus. A minimum of 14 days since the last dose of sirolimus is required prior to starting treatment with alpelisib
4. A documented genetic alteration in the PI3K signalling pathway identified by genetic sequencing prior to enrolment in this study
5. Adequate performance status (Eastern Cooperative Oncology Group Performance Status Scale (ECOG) 0-2 in patients ≥ 16 years of age; Lansky > 50 in patients < 16 years of age)
6. Patient has a life expectancy ≥ 12 weeks
7. Patient is able to swallow and retain oral medication
8. Adequate haematologic and end-organ function:

   * Haematology: Haemoglobin ≥ 9.0 g/dL; Absolute neutrophil count ≥ 1.5 x 109/L; Platelets ≥ 90 x 109/L, except where bleeding leading to low haemoglobin level is an indication for treatment, in which case haemoglobin < 9.0 g/dL is acceptable.
   * Hepatic function: alanine aminotransferase (ALT) and aspartate aminotransferase (AT) ≤ 3 x ULN; Total bilirubin < 2x ULN except for participants with Gilbert's syndrome who may only be included if the total bilirubin is ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN
   * Renal function: Serum creatinine < 1.5 x ULN
   * Biochemistry: Calcium (corrected for serum albumin) and magnesium within normal limits or ≤ Grade 1 according to NCI-CTCAE v5.0 if judged clinically not significant by the investigator; Potassium within normal limits, or corrected with supplements
   * Fasting blood glucose ≤ 7.0 mmol/L and Glycosylated Haemoglobin (HbA1c) ≤ 6.4% (both criteria must be met)
9. Patient agrees to abstinence or highly effective contraceptive measures for males and women of childbearing potential (WOCBP)

   * Males who are sexually active must use a condom during intercourse while taking alpelisib and for at least 4 weeks after stopping alpelisib and should not father a child in this period. A condom is required to be used also by vasectomised men in order to prevent delivery of the drug via seminal fluid. In addition, male participants must not donate sperm during the study and for at least 4 weeks after stopping alpelisib
   * Females who are of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use a highly effective method of contraception during study treatment and for at least 1 week after the last dose of any study treatment. Highly effective contraceptive methods include:

     * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject) Periodic abstinence (eg., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception;
     * Female sterilisation (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least 6 weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the women has been confirmed by follow up hormone level assessment;
     * Male partner sterilisation (at least 6 months prior to screening) of the sole partner of a female participant on the study;
     * Use of oral (estrogen and progesterone), injected or implanted combined hormonal method of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormonal vaginal ring or transdermal hormone contraception. In the case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
   * Women are considered postmenopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhoea with an appropriate clinical profile (i.e., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least 6 weeks before taking study treatment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered to be not of child bearing potential.
10. Patient has signed informed consent and is willing and able to comply with the protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations

Exclusion Criteria:

1. History of hypersensitivity to any drugs or metabolites of PI3K inhibitors or any of the excipients of alpelisib
2. Severe infection requiring intravenous antibiotics within 4 weeks prior to enrolment
3. Patient has had a major surgical procedure within 4 weeks prior to enrolment
4. Prior use of an alpha-specific PI3K inhibitor
5. History of pneumonitis or interstitial lung disease
6. Patient is pregnant or lactating at the time of study registration. A pregnancy test is mandated for women of child-bearing potential in the screening period
7. Established diagnosis of type I diabetes mellitus, type II diabetes mellitus requiring anti-hyperglycaemic medication or any participant with HbA1c > 6.4%
8. Patient who is currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes
9. Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to the start of treatment:

   * Strong inducers of CYP3A4
   * Strong inhibitors of CYP3A4
   * Inhibitors of BCRP
10. History of acute pancreatitis within 1 year of screening or past history of chronic pancreatitis
11. Patient with Child Pugh score B or C
12. Unresolved osteonecrosis of the jaw
13. Impairment of GI function or GI disease that may significantly alter the absorption of the study drug based on investigator discretion
14. Known history of Human Immunodeficiency Virus (HIV) infection (testing for HIV is not mandatory in screening)
15. Known history of severe cutaneous reactions like Stevens-Johnson Syndrome (SJS), Toxic Epidermal Necrolysis (TEN), Erythema Multiforme (EM), or Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS)
16. Known history of clinically significant, uncontrolled heart disease and/or recent cardiac events including:

    * History of angina pectoris, coronary artery bypass graft (CABG), symptomatic pericarditis, or myocardial infarction within 6 months prior to the start of study treatment;
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV);
    * History of impaired Left Ventricular Ejection Fraction (LVEF) < 50% (an assessment of LVEF is not mandatory in screening)
    * History of clinically significant cardiac arrhythmias, (e.g., ventricular tachycardia), complete left bundle branch block, high grade Atrioventricular (AV) block (e.g. bifascicular block, Mobitz type II and third degree AV block without pacemaker in place);
    * Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mmHg and/or Diastolic Blood Pressure (DBP) ≥ 100 mmHg, with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening;
    * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or corrected QT interval > 470 msec at screening (using Fridericia correction);
    * Bradycardia (heart rate < 50 beats per minute at rest), by electrocardiogram (ECG) or pulse
17. Patient has other concurrent severe and/or uncontrolled medical conditions that would, in the Treating Physician's judgement, contraindicate administration of alpelisib (eg. active or uncontrolled severe infection, chronic active hepatitis, immune-compromised, acute or chronic pancreatitis, uncontrolled high blood pressure)
18. Patient is unable to understand and comply with treatment instructions and requirements

MODULE 2

Inclusion Criteria:

1. Adult or paediatric patient, 2 years of age or over where Body Surface Area (BSA) is greater than or equal to 0.4m2.
2. Patient has a clinical diagnosis of a fast-flow vascular malformation
3. Patient has received standard therapy for the vascular malformation or in which, in the opinion of the investigator, standard therapy is not appropriate

   - Note: standard therapy may include treatment with sirolimus. A minimum of 14 days since the last dose of sirolimus is required prior to starting treatment with mirdametinib
4. A documented genetic alteration in the RAS-MEK-ERK signalling pathway identified by genetic sequencing prior to enrolment in this study
5. Adequate performance status (Eastern Cooperative Oncology Group Performance Status Scale (ECOG) 0-2 in patients ≥ 16 years of age; Lansky > 50 in patients < 16 years of age)
6. Patient has a life expectancy ≥ 12 weeks
7. Participant has the ability to swallow capsules whole if the capsule dosage form is being utilized. This criterion does not apply if participant is utilizing the dispersible tablet form of study treatment
8. Adequate haematologic and end-organ function:

   * Haematology: Haemoglobin ≥ 9.0 g/dL; Absolute neutrophil count ≥ 1.5 x 109/L; Platelets ≥ 90 x 109/L, except where bleeding leading to low haemoglobin level is an indication for treatment, in which case haemoglobin < 9.0 g/dL is acceptable.
   * Hepatic function: alanine aminotransferase (ALT) and aspartate aminotransferase (AT) ≤ 2 x upper limit of normal (ULN); Total bilirubin < 1.5x ULN (isolated bilirubin > 1.5x ULN is acceptable if bilirubin is fractioned and direct bilirubin < 35%), except where impaired hepatic function is a consequence of the fast-flow malformation and hence is an indication for treatment, in which case impaired hepatic function is acceptable.
   * Renal function: Serum creatinine < 1.5 x ULN
   * Biochemistry: Calcium (corrected for serum albumin) and magnesium within normal limits or ≤ Grade 1 according to NCI-CTCAE v5.0 if judged clinically not significant by the investigator; Potassium within normal limits or corrected with supplements; Phosphate ≤ 1x ULN.
9. Patient agrees to abstinence or highly effective contraceptive measures if of childbearing potential (WOCBP)

   * Males who are sexually active must use a condom during intercourse while taking mirdametinib and for at least 90 days after stopping mirdametinib and should not father a child in this period. A condom is required to be used also by vasectomised men in order to prevent delivery of the drug via seminal fluid. In addition, male participants must not donate sperm during the study and for at least 90 days after stopping mirdametinib
   * Females who are of child-bearing potential, defined as all individuals physiologically capable of becoming pregnant, must use a highly effective method of contraception during study treatment and for at least 180 days after the last dose of any study treatment. Highly effective contraceptive methods include:

     * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject) Periodic abstinence (eg., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception;
     * Female sterilisation (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least 6 weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the women has been confirmed by follow up hormone level assessment;
     * Male partner sterilisation (at least 6 months prior to screening) of the sole partner of a female participant on the study;
     * Use of oral (estrogen and progesterone), injected or implanted combined hormonal method of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormonal vaginal ring or transdermal hormone contraception. In the case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
   * Women are considered postmenopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhoea with an appropriate clinical profile (i.e., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least 6 weeks before taking study treatment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered to be not of childbearing potential.
10. Patient has signed informed consent and is willing and able to comply with the protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations

Exclusion Criteria:

1. History of hypersensitivity to any drugs or metabolites of MEK inhibitors or any of the excipients of mirdametinib
2. Severe infection requiring intravenous antibiotics within 4 weeks prior to enrolment
3. Patient has had a major surgical procedure within 4 weeks prior to enrolment
4. Prior use of a MEK inhibitor
5. Patient has abnormal QT interval corrected by Fridericia's formula (> 450 msec for male participants, > 470 msec for female participants, or > 480 msec for participants with bundle branch block) (triplicate ECG readings taken approximately 2 to 3 minutes apart and averaged) at Screening;
6. Patient is pregnant or lactating at the time of study registration. A pregnancy test is mandated for persons of child-bearing potential in the screening period
7. Impairment of GI function or GI disease that may significantly alter the absorption of the study drug based on investigator discretion
8. Any clinically significant active or known history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
9. Lymphoma, leukaemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years;
10. Breast cancer within the past 5 years;
11. Known history of Human Immunodeficiency Virus (HIV) infection (testing for HIV is not mandatory in screening)
12. Known history of severe cutaneous reactions like Stevens-Johnson Syndrome (SJS), Toxic Epidermal Necrolysis (TEN), Erythema Multiforme (EM), or Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS)
13. Patient has a history of, or evidence of, retinal pathology on ophthalmologic examination that is considered a risk factor for central serous retinopathy, retinal vein occlusion (RVO), or neovascular macular degeneration. Patients will be excluded from study participation if they have any of the following risk factors for RVO at Screening:

    * Intraocular pressure > 21 mmHg;
    * Serum cholesterol > 7.8 mmol/L;
    * Serum triglycerides > 3.4 mmol/L;
    * Hyperglycaemia (fasting blood glucose > 7.0 mol/L );
    * Age specific hypertension

      * Patients ≥ 13 years of age with a blood pressure ≥ 140/90 mmHg
      * Patients ≤ 12 years of age with a blood pressure ≥ 95th percentile for age + 12 mmHg
14. Known history of glaucoma
15. Known history of clinically significant, uncontrolled heart disease and/or recent (within 6 months [24 weeks] of signing informed consent/assent) cardiac events including:

    * History of angina pectoris, coronary artery bypass graft (CABG), symptomatic pericarditis, or myocardial infarction within 6 months prior to the start of study treatment;
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV);
    * History of clinically significant cardiac arrhythmias, (e.g., ventricular tachycardia), complete left bundle branch block, high grade Atrioventricular (AV) block (e.g. bifascicular block, Mobitz type II and third degree AV block without pacemaker in place);
    * Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 140 mmHg and/or Diastolic Blood Pressure (DBP) ≥ 90 mmHg, with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening;
    * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or corrected QT interval > 470 msec at screening (using Fridericia correction);
    * Bradycardia (heart rate < 50 beats per minute at rest), by electrocardiogram (ECG) or pulse
16. Patient has recorded a left ventricular ejection fraction (LVEF) < 55% at Screening
17. Patient has experienced a cerebrovascular accident, transient ischaemic attach, or symptomatic pulmonary embolism within 6 months (24 weeks) of signing informed consent/assent.
18. Patient has other concurrent severe and/or uncontrolled medical conditions that would, in the Treating Physician's judgement, contraindicate administration of mirdametinib (eg. active or uncontrolled severe infection, chronic active hepatitis, immune-compromised, acute or chronic pancreatitis, uncontrolled high blood pressure)
19. Patient is unable to understand and comply with treatment instructions and requirements

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The number of participants who achieve or exceed a predetermined threshold of improvement in their most significant symptom at 48 weeks based on the Vascular Malformation Patient Specific Outcome Measure (VM-PSOM). | At 48 weeks
  Vascular malformations present with a range of different symptoms. Therefore, there is no single outcome measure that can capture the effectiveness of a systemic treatment across different patients. Thus for this study, an individualised primary outcome for each patient informed by their symptoms will be used, termed the Vascular Malformation Patient Specific Outcome Measure (VM-PSOM). The study "Outcome Committee" will define an individualised primary outcome for each patient informed by their symptoms and vascular malformation features prior to starting trial treatments. The VM-PSOM endpoint will therefore define a binary outcome for each patients (achieved or failed to reach the threshold improvement in the chosen measure).

SECONDARY OUTCOMES:
The number of participants who achieve or exceed a predetermined threshold of improvement in their most significant symptom at the 168-day timepoint based on the Vascular Malformation Patient Specific Outcome Measure (VM-PSOM). | 48 weeks, 168-day follow-up
  VM-PSOM response at the 168 day follow-up visit assessment compared with the 48 week (end-of-treatment) VM-PSOM.
The number of participants with an objective response (defined as ≥ 20% reduction from index date in the sum of measurable target lesion volume) by volumetric analysis on MRI. | Baseline, 48 weeks
  Objective response rate by volumetric MRI assessment comparing 48 week (end-of-treatment) MRI with baseline MRI. MRI scan will only be performed in patients where their vascular malformation is feasibly evaluable by MRI scan. Objective response is defined as ≥ 20% reduction from index date in the sum of measurable target lesion volume by volumetric analysis on MRI.
Change in symptoms score as recorded on the OVAMA (Outcome measures for VAscular MAlformations) questionnaire. | Time frame: Baseline, 48 weeks
  The mean scores in the OVAMA (Outcome measures for VAscular MAlformations) questionnaire will be calculated and analysed at specified time points. This is a set of questions developed specifically to measure symptom burden from vascular malformations. These questions are open-ended to allow the subject to describe how they feel. The questions are more tightly structured to allow comparison of answers to other people with vascular malformations. The questions have been designed in a way to determine if symptoms are getting better over time.
Change in symptoms score as recorded on the OVAMA (Outcome measures for VAscular MAlformations) which is a set of questions developed specifically to measure symptom burden from vascular malformations. | Time frame: 48 weeks, Day 168 follow-up
  The mean scores in the OVAMA (Outcome measures for VAscular MAlformations) questionnaire will be calculated and analysed at specified time points.
The number of patients who experience adverse events as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5. | From Baseline to Day 168 follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Tony Penington, MBBS, FRACS., Principal Investigator — Study Principal Investigator; Stephen Luen, MBChB, FRACP., Principal Investigator — Principal Investigator; Lydia Pathmanathan, MBBS, FRACP., Principal Investigator — Principal Investigator
Locations (2):
- Australia (2):
  - Peter MacCallum Cancer Centre, Parkville, Victoria
  - The Royal Children's Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: Yes
From 6 months post analysis and article publication, the following will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept The Murdoch Children's Research Institute's (MCRI) conditions for access:
  * Individual participant data that underlie the results reported in this article after de-identification
  * Trial protocol, Statistical Analysis Plan, PICF The Sponsor-Investigator will be the long-term custodian after the archive period has finished.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available from 6 months following analysis and article publication
Access Criteria: Future researchers must be from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access

REFERENCES:
- [Background] Garzon MC, Huang JT, Enjolras O, Frieden IJ. Vascular malformations: Part I. J Am Acad Dermatol. 2007 Mar;56(3):353-70; quiz 371-4. doi: 10.1016/j.jaad.2006.05.069. PMID 17317485
- [Background] Penington, A.P., R.; Sleebs, N.; Halliday, J. , Epidemiology of Vascular Malformations Poster, in International Society for the Study of Vascluar Anomalies World Congress. 2022: Vancouver, British Columbia, Canada.
- [Background] Wagner KM, Lokmic Z, Penington AJ. Prolonged antibiotic treatment for infected low flow vascular malformations. J Pediatr Surg. 2018 Apr;53(4):798-801. doi: 10.1016/j.jpedsurg.2017.05.022. Epub 2017 May 27. PMID 28599969
- [Background] Cheng J, Liu B, Farjat AE, Routh J. The Public Health Burden of Lymphatic Malformations in Children: National Estimates in the United States, 2000-2009. Lymphat Res Biol. 2017 Sep;15(3):241-245. doi: 10.1089/lrb.2017.0009. Epub 2017 Jul 31. PMID 28759318
- [Background] Liu AS, Mulliken JB, Zurakowski D, Fishman SJ, Greene AK. Extracranial arteriovenous malformations: natural progression and recurrence after treatment. Plast Reconstr Surg. 2010 Apr;125(4):1185-1194. doi: 10.1097/PRS.0b013e3181d18070. PMID 20335868
- [Background] Chen RJ, Vrazas JI, Penington AJ. Surgical Management of Intramuscular Venous Malformations. J Pediatr Orthop. 2021 Jan;41(1):e67-e73. doi: 10.1097/BPO.0000000000001667. PMID 32815867
- [Background] Leaute-Labreze C, Dumas de la Roque E, Hubiche T, Boralevi F, Thambo JB, Taieb A. Propranolol for severe hemangiomas of infancy. N Engl J Med. 2008 Jun 12;358(24):2649-51. doi: 10.1056/NEJMc0708819. No abstract available. PMID 18550886
- [Background] Hammill AM, Wentzel M, Gupta A, Nelson S, Lucky A, Elluru R, Dasgupta R, Azizkhan RG, Adams DM. Sirolimus for the treatment of complicated vascular anomalies in children. Pediatr Blood Cancer. 2011 Dec 1;57(6):1018-24. doi: 10.1002/pbc.23124. Epub 2011 Mar 28. PMID 21445948
- [Background] Adams DM, Trenor CC 3rd, Hammill AM, Vinks AA, Patel MN, Chaudry G, Wentzel MS, Mobberley-Schuman PS, Campbell LM, Brookbank C, Gupta A, Chute C, Eile J, McKenna J, Merrow AC, Fei L, Hornung L, Seid M, Dasgupta AR, Dickie BH, Elluru RG, Lucky AW, Weiss B, Azizkhan RG. Efficacy and Safety of Sirolimus in the Treatment of Complicated Vascular Anomalies. Pediatrics. 2016 Feb;137(2):e20153257. doi: 10.1542/peds.2015-3257. Epub 2016 Jan 18. PMID 26783326
- [Background] Hammer J, Seront E, Duez S, Dupont S, Van Damme A, Schmitz S, Hoyoux C, Chopinet C, Clapuyt P, Hammer F, Vikkula M, Boon LM. Sirolimus is efficacious in treatment for extensive and/or complex slow-flow vascular malformations: a monocentric prospective phase II study. Orphanet J Rare Dis. 2018 Oct 29;13(1):191. doi: 10.1186/s13023-018-0934-z. PMID 30373605
- [Background] Keppler-Noreuil KM, Sapp JC, Lindhurst MJ, Parker VE, Blumhorst C, Darling T, Tosi LL, Huson SM, Whitehouse RW, Jakkula E, Grant I, Balasubramanian M, Chandler KE, Fraser JL, Gucev Z, Crow YJ, Brennan LM, Clark R, Sellars EA, Pena LD, Krishnamurty V, Shuen A, Braverman N, Cunningham ML, Sutton VR, Tasic V, Graham JM Jr, Geer J Jr, Henderson A, Semple RK, Biesecker LG. Clinical delineation and natural history of the PIK3CA-related overgrowth spectrum. Am J Med Genet A. 2014 Jul;164A(7):1713-33. doi: 10.1002/ajmg.a.36552. Epub 2014 Apr 29. PMID 24782230
- [Background] Venot Q, Blanc T, Rabia SH, Berteloot L, Ladraa S, Duong JP, Blanc E, Johnson SC, Hoguin C, Boccara O, Sarnacki S, Boddaert N, Pannier S, Martinez F, Magassa S, Yamaguchi J, Knebelmann B, Merville P, Grenier N, Joly D, Cormier-Daire V, Michot C, Bole-Feysot C, Picard A, Soupre V, Lyonnet S, Sadoine J, Slimani L, Chaussain C, Laroche-Raynaud C, Guibaud L, Broissand C, Amiel J, Legendre C, Terzi F, Canaud G. Targeted therapy in patients with PIK3CA-related overgrowth syndrome. Nature. 2018 Jun;558(7711):540-546. doi: 10.1038/s41586-018-0217-9. Epub 2018 Jun 13. PMID 29899452
- [Background] Canaud, G., et al., LBA23 EPIK-P1: Retrospective chart review study of patients (pts) with PIK3CA-related Overgrowth Spectrum (PROS) who have received alpelisib (ALP) as part of a compassionate use programme. Annals of Oncology, 2021. 32: p. S1297.
- [Background] Al-Olabi L, Polubothu S, Dowsett K, Andrews KA, Stadnik P, Joseph AP, Knox R, Pittman A, Clark G, Baird W, Bulstrode N, Glover M, Gordon K, Hargrave D, Huson SM, Jacques TS, James G, Kondolf H, Kangesu L, Keppler-Noreuil KM, Khan A, Lindhurst MJ, Lipson M, Mansour S, O'Hara J, Mahon C, Mosica A, Moss C, Murthy A, Ong J, Parker VE, Riviere JB, Sapp JC, Sebire NJ, Shah R, Sivakumar B, Thomas A, Virasami A, Waelchli R, Zeng Z, Biesecker LG, Barnacle A, Topf M, Semple RK, Patton EE, Kinsler VA. Mosaic RAS/MAPK variants cause sporadic vascular malformations which respond to targeted therapy. J Clin Invest. 2018 Apr 2;128(4):1496-1508. doi: 10.1172/JCI98589. Epub 2018 Mar 12. PMID 29461977
- [Background] Dombi E, Ardern-Holmes SL, Babovic-Vuksanovic D, Barker FG, Connor S, Evans DG, Fisher MJ, Goutagny S, Harris GJ, Jaramillo D, Karajannis MA, Korf BR, Mautner V, Plotkin SR, Poussaint TY, Robertson K, Shih CS, Widemann BC; REiNS International Collaboration. Recommendations for imaging tumor response in neurofibromatosis clinical trials. Neurology. 2013 Nov 19;81(21 Suppl 1):S33-40. doi: 10.1212/01.wnl.0000435744.57038.af. PMID 24249804
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Matthews HS, Penington AJ, Hardiman R, Fan Y, Clement JG, Kilpatrick NM, Claes PD. Modelling 3D craniofacial growth trajectories for population comparison and classification illustrated using sex-differences. Sci Rep. 2018 Mar 19;8(1):4771. doi: 10.1038/s41598-018-22752-5. PMID 29556038
- [Background] Fan Y, Penington A, Kilpatrick N, Hardiman R, Schneider P, Clement J, Claes P, Matthews H. Quantification of mandibular sexual dimorphism during adolescence. J Anat. 2019 May;234(5):709-717. doi: 10.1111/joa.12949. Epub 2019 Mar 4. PMID 30834524
- [Background] Turk DC, Dworkin RH, Allen RR, Bellamy N, Brandenburg N, Carr DB, Cleeland C, Dionne R, Farrar JT, Galer BS, Hewitt DJ, Jadad AR, Katz NP, Kramer LD, Manning DC, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robinson JP, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Witter J. Core outcome domains for chronic pain clinical trials: IMMPACT recommendations. Pain. 2003 Dec;106(3):337-345. doi: 10.1016/j.pain.2003.08.001. PMID 14659516
- [Background] Patel KV, Amtmann D, Jensen MP, Smith SM, Veasley C, Turk DC. Clinical outcome assessment in clinical trials of chronic pain treatments. Pain Rep. 2021 Jan 21;6(1):e784. doi: 10.1097/PR9.0000000000000784. eCollection 2021 Jan-Feb. PMID 33521482
- [Background] Stinson JN, Kavanagh T, Yamada J, Gill N, Stevens B. Systematic review of the psychometric properties, interpretability and feasibility of self-report pain intensity measures for use in clinical trials in children and adolescents. Pain. 2006 Nov;125(1-2):143-57. doi: 10.1016/j.pain.2006.05.006. Epub 2006 Jun 13. PMID 16777328
- [Background] Younger J, McCue R, Mackey S. Pain outcomes: a brief review of instruments and techniques. Curr Pain Headache Rep. 2009 Feb;13(1):39-43. doi: 10.1007/s11916-009-0009-x. PMID 19126370
- [Background] Smith SM, Dworkin RH, Turk DC, McDermott MP, Eccleston C, Farrar JT, Rowbotham MC, Bhagwagar Z, Burke LB, Cowan P, Ellenberg SS, Evans SR, Freeman RL, Garrison LP, Iyengar S, Jadad A, Jensen MP, Junor R, Kamp C, Katz NP, Kesslak JP, Kopecky EA, Lissin D, Markman JD, Mease PJ, O'Connor AB, Patel KV, Raja SN, Sampaio C, Schoenfeld D, Singh J, Steigerwald I, Strand V, Tive LA, Tobias J, Wasan AD, Wilson HD. Interpretation of chronic pain clinical trial outcomes: IMMPACT recommended considerations. Pain. 2020 Nov;161(11):2446-2461. doi: 10.1097/j.pain.0000000000001952. PMID 32520773
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Fritsch C, Huang A, Chatenay-Rivauday C, Schnell C, Reddy A, Liu M, Kauffmann A, Guthy D, Erdmann D, De Pover A, Furet P, Gao H, Ferretti S, Wang Y, Trappe J, Brachmann SM, Maira SM, Wilson C, Boehm M, Garcia-Echeverria C, Chene P, Wiesmann M, Cozens R, Lehar J, Schlegel R, Caravatti G, Hofmann F, Sellers WR. Characterization of the novel and specific PI3Kalpha inhibitor NVP-BYL719 and development of the patient stratification strategy for clinical trials. Mol Cancer Ther. 2014 May;13(5):1117-29. doi: 10.1158/1535-7163.MCT-13-0865. Epub 2014 Mar 7. PMID 24608574
- [Background] Janku F, Hong DS, Fu S, Piha-Paul SA, Naing A, Falchook GS, Tsimberidou AM, Stepanek VM, Moulder SL, Lee JJ, Luthra R, Zinner RG, Broaddus RR, Wheler JJ, Kurzrock R. Assessing PIK3CA and PTEN in early-phase trials with PI3K/AKT/mTOR inhibitors. Cell Rep. 2014 Jan 30;6(2):377-87. doi: 10.1016/j.celrep.2013.12.035. Epub 2014 Jan 16. PMID 24440717
- [Background] Anderson NG, Maller JL, Tonks NK, Sturgill TW. Requirement for integration of signals from two distinct phosphorylation pathways for activation of MAP kinase. Nature. 1990 Feb 15;343(6259):651-3. doi: 10.1038/343651a0. PMID 2154696
- [Background] Roskoski R Jr. ERK1/2 MAP kinases: structure, function, and regulation. Pharmacol Res. 2012 Aug;66(2):105-43. doi: 10.1016/j.phrs.2012.04.005. Epub 2012 Apr 27. PMID 22569528
- [Background] Hoshino R, Chatani Y, Yamori T, Tsuruo T, Oka H, Yoshida O, Shimada Y, Ari-i S, Wada H, Fujimoto J, Kohno M. Constitutive activation of the 41-/43-kDa mitogen-activated protein kinase signaling pathway in human tumors. Oncogene. 1999 Jan 21;18(3):813-22. doi: 10.1038/sj.onc.1202367. PMID 9989833
- [Background] Weiss BD, Wolters PL, Plotkin SR, Widemann BC, Tonsgard JH, Blakeley J, Allen JC, Schorry E, Korf B, Robison NJ, Goldman S, Vinks AA, Emoto C, Fukuda T, Robinson CT, Cutter G, Edwards L, Dombi E, Ratner N, Packer R, Fisher MJ. NF106: A Neurofibromatosis Clinical Trials Consortium Phase II Trial of the MEK Inhibitor Mirdametinib (PD-0325901) in Adolescents and Adults With NF1-Related Plexiform Neurofibromas. J Clin Oncol. 2021 Mar 1;39(7):797-806. doi: 10.1200/JCO.20.02220. Epub 2021 Jan 28. PMID 33507822